CLINICAL TRIAL: NCT05903599
Title: Effects of Anodal Transcranial Direct Current Stimulation on Postural Stability in Sub-Acute Stroke
Brief Title: Anodal TDCS and Postural Stability in Subacute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC01353 Somia Shakeb
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): anodal Transcranial direct current stimulation with saline soaked sponges will be used on electrodes, for 20 mins in addition to the 60 mins of conventional treatment.
  Interventions: Other: Anodal transcranial direct current stimulation
- Group B (Sham Comparator): A sham stimulation will be given. It will be comprised 20 min of sham TDCS followed by 60 mins of conventional treatment for postural stability in sub-acute stroke
  Interventions: Other: Sham Stimulation

INTERVENTIONS:
Other: Anodal transcranial direct current stimulation — The size of both electrodes will be 5cm x 5cm placed on the head with the anode on the primary motor cortex M1 of the affected side while the cathode on the contralesional eye. The duration of the stimulation of anodal TDCS is 20 min and the intensity of current will be 2mA. The ramp up and down period will be 30se each. Treatment duration will be 5 times a week for 6 weeks for postural stability.
  Arms: Group A
Other: Sham Stimulation — postural training by visual feedback and weight shifting towards the non-paretic side. This program will have two phases. Phase one have 4 stages; The first stage (sessions 1-7), second stage (sessions 8-14), third stage (sessions 15-22), fourth stage (sessions 23-30).
  Next phase will include the exercises including balancing exercises.
  Arms: Group B

SUMMARY:
Stroke patients experience weakening of muscles on the affected side. Damage to the motor cortex and the pyramidal tract due to a stroke leads to a motor control disorders and co-contraction of trunk muscles due to abnormal levels of abdominal muscle tension and voluntary movement.

DETAILED DESCRIPTION:
TDCS is known to modulate motor excitability in humans and motor performance is crucial in postural control. Studies reports that applying anodal TDCS to the ipsilesional motor cortex improved motor functioning in which the Transcranial Direct Current Stimulation may have stimulated preserved areas of the motor cortex to enhance synaptic efficiency along the corticospinal tract.

Anodal TDCS has been shown to have immediate and short-term effects in stroke but its long-term effects in stroke are still unclear. Additionally, the available literature focuses on acute and chronic stages of stroke so we will target subacute stage of stroke. Therefore, this study is designed to investigate the short and long-term effects of Anodal Transcranial Direct Current Stimulation on postural stability in subacute stroke.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke
* Sub-acute stroke
* Minimum score of 18 on PASS

Exclusion Criteria:

Hearing and Visual loss/ deficit

* Recurrent CVA
* Neurological condition affects the cognition
* Wound at skull
* Presence of shunt and/or metallic implant at cranial region
* Brain tumors
* Musculoskeletal conditions/ surgery in the lower extremities
* Cognitively compromised

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Postural Assessment Scale for Stroke Patients (PASS) | 12th week
  PASS evaluates the postural imbalance and functional abilities of patients with stroke in several conditions (lying on back, sitting, standing and while changing positions). This scale is composed of 12 items. Score can vary from 0 to 3, with 0 being the lowest level of functionality and 3 the highest; the total score be 36.
Trunk impairment scale (TIS) for Stroke Patients | 12th week
  It evaluates motor impairment of the trunk after stroke. The TIS scores, on a range from 0 to 23, static and dynamic sitting trunkal stability as well as trunk coordination. It also score the quality of trunk movement and to be a guide for treatment. Number of items are 7, score of each item is 0-3.

SECONDARY OUTCOMES:
Timed Up and Go Test (TUG) | 12th week
  TUG test is a general performance test used to assess mobility, balance and locomotor performance in patients with balance disturbances. The patients are asked to stand up from chair, walk to a line of 3 meters length at a normal pace, turn and walk back to the chair at your normal pace and sit down. A patient whose score is less than 10 seconds is characterized as completely independent. Assessment time will be at 0, 3rd, 6th,9th,12th week
Functional Reach Test (FRT) | 12th week
  a clinical outcome measure and assessment tool for ascertaining dynamic balance in one simple task. The patient is instructed to stand next to but not touching a wall and position the arm that is closer to the wall at 90 degrees of shoulder flexion with a closed fist. The assessor records the starting position at the third metacarpal head on the yardstick. Instruct the patient to reach as far as you can forward without taking a step. The location of the third metacarpal is recorded. Scores are determined by assessing the difference between the start and end positions in the reach distance usually measured in inches. Three trials should be done and the average of the last two is noted. Assessment time will be at 0, 3rd, 6th,9th,12th week
Stroke Specific Quality of life Scale (SS-QoL) | 12th week
  a reliable and valid tool for measuring self-reported health -related quality of life. It is a patient centered outcome measure intended to provide an assessment of health-related quality of life specific with stroke. Scale domains and items were derived from series of interviews with post stroke patients. They must respond to each question of the SS-QOL with reference to the past week. It contains 49 items in 12 domains: mobility, energy, upper extremity function (5 items), work/productivity (3 items ), mood (5 items), social roles (5 items),family roles (3 items ), language (5 items ), thinking (3 items), personality (3 items) higher scores indicate better functioning. Assessment time will be at 0, 3rd, 6th,9th,12th week

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saeys W, Vereeck L, Lafosse C, Truijen S, Wuyts FL, Van De Heyning P. Transcranial direct current stimulation in the recovery of postural control after stroke: a pilot study. Disabil Rehabil. 2015;37(20):1857-63. doi: 10.3109/09638288.2014.982834. Epub 2015 Jul 9. PMID 25401406
- [Background] Halmi Z, Stone TW, Dinya E, Mally J. Postural instability years after stroke. J Stroke Cerebrovasc Dis. 2020 Sep;29(9):105038. doi: 10.1016/j.jstrokecerebrovasdis.2020.105038. Epub 2020 Jun 23. PMID 32807450
- [Background] Bornheim S, Croisier JL, Maquet P, Kaux JF. Transcranial direct current stimulation associated with physical-therapy in acute stroke patients - A randomized, triple blind, sham-controlled study. Brain Stimul. 2020 Mar-Apr;13(2):329-336. doi: 10.1016/j.brs.2019.10.019. Epub 2019 Oct 31. PMID 31735645